CLINICAL TRIAL: NCT05673096
Title: Paediatric Autism Communication Therapy (PACT) Combined With Management as Usual Compared to Management as Usual Alone in Children With Autism Spectrum Disorder - a Pragmatic, National, Randomised Clinical Trial
Brief Title: Paediatric Autism Communication Therapy (PACT) in Children With Autism Spectrum Disorder
Acronym: DAN-PACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); Region Capital Denmark (Other); Region Zealand (Other); Region of Southern Denmark (Other); Central Denmark Region (Other); Regionshospital Nordjylland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAN-PACT
Record Dates: First submitted 2022-12-22; First posted 2023-01-06 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the intervention, blinding of parents and therapists is impossible. The primary outcome measure, Autism Diagnostic Observation Schedule, Calibrated Severity Score (ADOS-CSS), and further outcomes (Brief Observation of Social Communication Change (BOSCC), Dyadic Communication Measure for Autism (DCMA) and Measure of Naturalistic Developmental Behavioral Intervention Strategy Implementation - Caregiver Change (MONSI-CC)) are videotaped, leaving raters blinded to treatment allocation. At the clinical follow-up assessment, families are asked not to reveal group allocation.
  Data from the DAN-PACT trial will be kept separate from research data and will not be accessible to the research team. We will follow the rule that statistical analyses are conducted with the intervention groups coded. The steering committee will write two abstracts while the blinding is intact assuming either group as intervention group and control, respectively. After this, the code will be broken
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PACT + Management as usual (Experimental): PACT + management (MAU - see comparator intervention). PACT is a parent-mediated and video-aided intervention designed to improve socio-communicative functioning in children with ASD. The intervention is based on theory and research on pre-linguistic and early social interaction and language development. The programme focuses on changing the interaction in the parent-child dyad in order to enhance communication and language development and skills in children with ASD.
  The overall focus of the intervention is to guide parents to provide a sensitive, highly adapted interaction context in which their own responses and language are matched to the child's communication competence and language comprehension. Parents learn to identify windows of opportunity to facilitate joint interactions, enhance emerging communication, elicit child intentionality and support language comprehension, thereby aiming to ameliorate abnormal developmental pathways.
  Interventions: Behavioral: PACT
- Management as usual (Active Comparator): Enhanced management as usual (MAU). MAU is delivered by the regional Child and Adolescent Mental Health Center (CAMHS). All participants will have equal access to seek advice via a telephone hotline in the trial period (12 months).
  Following the diagnosis of ASD, the parents will be offered psychoeducation as usual in the local CAMHS. A telephone "hotline" open to all participants will offer pedagogical advice and try to help the parents to collaborate and engage with their professional partners in the municipality. The parents will also be able to contact the CAMHS when needed. The hotline team will be able to consult with the responsible clinician at the CAMHS. The clinician should always be notified within the same day, if a parent describes acute worsening of the child's condition, risk of suicidality, or severe aggression. The responsible clinician will be able to refer the child to further assessment and treatment within the CAMHS without any significant delay.
  Interventions: Behavioral: MAU

INTERVENTIONS:
Behavioral: PACT — Paediatric Autism Communication Therapy
  Arms: PACT + Management as usual
Behavioral: MAU — Management as usual
  Arms: Management as usual

SUMMARY:
Paediatric Autism Communication Therapy (PACT) is a naturalistic developmental behavioural interventions to reduce autism symptoms. The aim of this trial is to assess the beneficial and harmful effects of PACT in 2-6 year-old children with a recent diagnosis of autism spectrum disorder.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a neurodevelopmental disorder affecting approximately 2% of children and young people worldwide. ASD is considered a lifelong disorder and interventions significantly reducing the core autistic symptoms have been sparse. Paediatric Autism Communication Therapy (PACT) is among the first naturalistic developmental behavioural interventions to show promising results for reduction in autism symptoms.

The aim of this trial is to assess the beneficial and harmful effects of PACT in 2-6 year-old children with a recent diagnosis of ASD.

This trial is an investigator-initiated, independently funded, pragmatic, national, parallel group, superiority, randomised clinical trial comparing PACT combined with management as usual to management as usual alone.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 through 6 years (both inclusive)
* A diagnosis of ASD meeting the criteria for International Classification of Diseases; Tenth Edition (ICD-10): Diagnose codes: DF84.0, DF84.1, DF84.5, DF84.8
* An Autism Diagnostic Observation Schedule, 2nd Edition Calibrated Severity Score (ADOS-2 CSS) ≥ 4
* The ASD diagnosis must be verified by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), Autism Spectrum Disorder Checklist
* The ASD diagnosis must be the primary developmental disorder (comorbid conditions allowed) and conferred at a clinical conference
* Parents must have sufficient Danish (or English) language skills to communicate with the therapist
* Signed informed consent by parents or holders of legal guardianship

Exclusion Criteria:

* Children having a sibling already included in the trial
* Hearing and visual impairment in child or parent
* Parent not available for regular sessions with the therapist, evaluated at the consent meeting

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 280 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Autism Symptoms | End of intervention (14 months)
  Autism symptoms are measured by Diagnostic Observation schedule, 2nd Edition, Calibrated Severity Score (ADOS-2 CSS). Range 0-10, with 10 indicating the highest symptom severity.

SECONDARY OUTCOMES:
Child adaptive functioning | End of intervention (14 months)
  Child adaptive functioning, or personal and social skills needed for everyday living will be measured by the Vineland Adaptive Behavior Scales, 3rd Edition (VABS-3), an online questionnaire filled in by parents. Each of four domains, Communication, Daily Living Skills, Socialization and Motor Skills are divided into 3 sub-domains. Each item is scored on a Likert-type format with scores 0 (never), 1(sometimes), and 2 (usually or often). Individual items scores are summed to a raw composite score and converted into a standard scale scores. Higher scores indicate higher functioning.
Social interaction of the child | At 6 month and end of intervention (14 months)
  Brief Observation of Social Communication Change (BOSCC) is rated on a 12-minute videotaped parent-child play-session. Each of the 15 behavioural items is coded using an empirically based decision tree that captures information regarding the behaviour including frequency and quality. Each item is rated on a 6- point scale from 0 (abnormality is not present) to 5 (abnormality is present and significantly impairs functioning). For measuring change only item 1-12 (range 0-60) are used.
Quality of Life (child) | End of intervention (14 months)
  Parents' assessment of their child's quality of life with Pediatric Quality of Life Inventory (PEDSQL), a questionnaire including 23 items covering four dimensions of health related quality of life. Each item is rated between 0 and 100. A higher score indicates a higher level of health-related quality of life. The mean item score is used as outcome.
Quality of life (parents) | End of intervention (14 months)
  Parent quality of life is measured by the questionnaire World Health Organization Quality of Life assessment- BREF (WHOQOL-BREF), including 28 items of quality of life for parents in 4 dimensions: Physiological, emotional, social and context. The item scores range from 1 to 5 with higher scores denoting higher quality of life. As the number of items differs for each subscale, the mean item score is used as outcome.

OTHER OUTCOMES:
Parent-child synchrony and initiative in communication | At 6 month and end of intervention (14 months)
  Dyadic Communication Measure for Autism (DCMA) is used to rate parent synchrony and responsiveness to the child, child communicative initiations, responses and communicative functions, and amount of mutual shared attention between parent and child will be measured by the DCMA. DCMA is rated on a 12-minute videotaped parent-child play-session. Raters will be blinded to treatment allocation.
Parent implementation of strategy | End of intervention (14 months)
  Caregivers' implementation of PACT strategies will be measured by the Measure of Naturalistic Developmental Behavioral Intervention Strategy Implementation - Caregiver Change (MONSI-CC) rated on a 12-minute videotaped parent-child play-session. Each of 21 items are rated between 1 (strategy was rarely implemented) and 5 (strategies were well-timed) and summed on different subscales. Raters will be blinded to treatment allocation.
Behavioural and emotional problems | End of intervention (14 months)
  Child symptoms and problems are measured by the Child Behavior Checklist for ages 1½-5 (CBCL/1½-5). A 99 item questionnaire generating a Total problem Score (range 0-198). Higher score indicating more problems
Family life functioning | End of intervention (14 months)
  Participant family life functioning will be measured by the Autism Family Experience Questionnaire (AFEQ). A parent-reported questionnaire with 48 items (range 48-240). High score indication low function.
Social impairment | End of intervention (14 months)
  The presence and severity of social impairment will be measured by the Social Responsiveness Scale, 2nd Edition (SRS-2). A parent reported questionnaire with 65 items identifying the presence and severity of social impairment. Each item is scored on a 4 point Likert-scale: 1 ("not true"); 2 ("sometimes true); 3 (often true); and 4 ("almost always true"). Scores are obtained for five Treatment Subscales: Social Awareness; Social Cognition; Social Communication; Social Motivation; and Restricted Interests and Repetitive Behavior. Higher scores indicating more severe impairment.
Parental reflective functioning | End of intervention (12 months)
  Parental reflective functioning will be measured by the Parental Reflective Functioning Questionnaire (PRFQ-1) with 18 items all rated on a 7-point scale with (7 if you strongly agree; and 1 if you strongly disagree. The midpoint, if you are neutral or undecided, is 4). High score indicate highly or hyper- reflective
Child attachment | End of intervention (14 months)
  Parents' perception of their child's attachment is rated on the Maternal Perception of Child Attachment (MPCA). This parent-report measure consists of 23 items rated on a 5-point rating scale, ranging from frequently (1) to never (5). High scores indicate maternal perceptions of strong child attachment.
Adverse events | End of intervention (14 months)
  Adverse events that occur during the study will be measured by the Negative Effects Questionnaire (NEQ). The NEQ questionnaire measures six factors; symptoms, quality, dependency, stigma, hopelessness, and failure. The self-report measure consists of three parts. First, respondents endorse specific items in case they have occurred or not during treatment, yes/no (1/0). Second, the respondents rate how negatively the negative effect was on four-point Likert-scale, ranging from "Not at all" to "Extremely" (0-4). Third, the respondents attribute the negative effect to "The treatment I received" yes/no (1/0).
Serious Adverse Events | End of intervention (14 months)
  Serious Adverse Events (SAE) defined as any adverse event (AE) that results in death, is life-threatening, requires hospitalisation or prolongation of existing hospitalisation, or results in persistent or significant disability or incapacity is registered continuously through patient files
Cost-effectiveness | End of intervention (14 months)
  The costs of delivering PACT combined with MAU compared to MAU alone will be estimated through cost-effectiveness analyses of intervention deliveries and parents' productivity loss
Parents' perceptions of the intervention | End of intervention (14 months)
  Parents' perceptions of the intervention will be explored in a subsample of parents in each intervention group by qualitative interviews
Receptive language | End of intervention (14 months)
  Child receptive language as measured by the Mullens Scales of Early Learning (MSEL). The MSEL consists of four cognitive scales: Visual Reception, Fine Motor, Receptive Language, Expressive Language, as well as a Gross Motor Scale, and can be administered to infants and children up to 5 years, 6 months of age. The MSEL receptive language raw scores will be used for the total study population in order to use the same instrument for all children, even when some of them may be older than the validated target group.
Language | End of intervention (14 months)
  Child language as measured by the New Reynell Developmental Language Scale (NRDLS). The NRDLS covers a number of important aspects of language acquisition including vocabulary, sentence structure, verb morphology, inference, and grammaticality judgement. NRDLS is developed for children 2-7 years of age. The NRDLS raw scores will be used for the total study population in order to use the same instrument for all children, even when some of them may older than the validated target group at follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Bilenberg, Professor, Study Chair — Department of Child and Adolescent Mental Health Odense, Mental Health Services in the Region of Southern Denmark + Clinical Institute, University of Southern Denmark
Locations (6):
- Denmark (6):
  - Child and Adolescent Mental Health Center, Aabenraa, Region of Southern Denmark, Aabenraa
  - Child and Adolescent Mental Health Center, Aalborg, North Denmark Region, Aalborg
  - Child and Adolescent Psychiatric Dept., Skejby, Aarhus University Hospital, Aarhus
  - Child and Adolescent Mental Health Center, Capital Region of Denmark, Hellerup
  - Child and Adolescent Mental Health Center, Odense, Region of Southern Denmark, Odense
  - Department of Child and Adolescent Psychiatry, Copenhagen University Hospital, Roskilde

IPD SHARING:
Plan to Share IPD: Yes
After the results have been published, we aim to make a depersonalized dataset publicly available on e.g. clinicaltrials.gov and/or the European Union (EU) Zenodo database. The final choice will reflect which platform(s) that are compliant with current legislation at that time.
Supporting Information: Study Protocol, SAP
Time Frame: When the results have been published
Access Criteria: Researchers with a protocol for their planned study

REFERENCES:
- [Derived] Ziegler SMT, Jeppesen P, Christiansen J, Conrad CE, Davidsen KA, Engkjaer-Trautwein G, Engstrom J, Fagerlund B, Gotzsche MV, Hastrup LH, Jakobsen JC, Kirk AM, Lauritsen MB, Pagsberg AK, Pedersen MA, Kilburn TR, Thomsen PH, Varenne M, Bilenberg N. Paediatric Autism Communication Therapy (PACT) versus management as usual in autistic children: a protocol for a Danish pragmatic, national, randomised clinical trial: DAN-PACT. Trials. 2025 Aug 29;26(1):322. doi: 10.1186/s13063-025-09017-z. PMID 40883837